CLINICAL TRIAL: NCT01266889
Title: Measurement of Cerebral Oxygenation Using NIRS Method in the Preterm Infants With Intracranial Haemorrhagia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Zekai Tahir Burak Maternity and Teaching Hospital, Zekai Tahir Burak Maternity and Teaching Hospital
Other Study IDs: 3
Record Dates: First submitted 2010-12-06; First posted 2010-12-24 (Estimated); Last update posted 2010-12-24 (Estimated); Status verified 2010-12

CONDITIONS: Cerebral Oxygenation, Intracranial Haemorrhagia
Keywords: preterm infant,cerebral oxygenation, intracranial haemorrhagia
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- study group, control group
  Interventions: Device: device:INVOS 5100

INTERVENTIONS:
Device: device:INVOS 5100 — Continuous wave NIRS is a method for measurement of cerebral oxygenation and haemodynamics. This method is non-invasive, continuous, and can also be used as bedside monitoring. With continuous wave NIRS only changes in concentration of oxyhaemoglobin (O2Hb) and deoxyhaemoglobin (HHb) can be measured, not the absolute level of these parameters. It has been shown that changes in concentration of HbD (O2Hb - HHb) reflect changes in CBF. So, continuous monitoring of changes in concentration of HbD can be used as an indicator of changes in CBF, but changes in CBV will also influence the HbD signal, as will changes in arterial O2 saturation (saO2) and changes in cerebral metabolic rate for oxygen.

SUMMARY:
The aim of the study was investigated the cerebral tissue oxygenation index (c-TOI) measured by near infrared spectroscopy (NIRS)in the preterm infants with intracranial haemorrhagia.

ELIGIBILITY:
Inclusion Criteria:

.<34 gestation week preterm infants with intracranial haemorrhagia

Exclusion Criteria:

* sepsis
* NEC
* congenital abnormalities
* hydrocephalus
* intracranial infections

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: primer care clinic
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-03 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
cerebral oxygenation | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Melek Akar, Ankara, Hamamönü, Turkey (Türkiye)